CLINICAL TRIAL: NCT01578707
Title: A Randomized, Multicenter, Open-label, Phase 3 Study of the Bruton's Tyrosine Kinase (BTK) Inhibitor Ibrutinib (PCI-32765) Versus Ofatumumab in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: A Phase 3 Study of Ibrutinib (PCI-32765) Versus Ofatumumab in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia
Acronym: RESONATE™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1112-CA; 2012-000694-23 (EudraCT Number)
Record Dates: First submitted 2012-04-11; First posted 2012-04-17 (Estimated); Results first posted 2015-10-12 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Relapsed or Refractory Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Chronic; SLL; CLL; Ofatumumab; ibrutinib; RESONATE; Phase III; Leukemia; Lymphoma
MeSH Terms: conditions — Recurrence; Leukemia, Lymphocytic, Chronic, B-Cell; Bronchiolitis Obliterans Syndrome; Leukemia; Lymphoma | interventions — ofatumumab; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ofatumumab (Arm A) (Active Comparator): An anti-CD20 monoclonal antibody
  Interventions: Drug: ofatumumab
- ibrutinib (Arm B) (Experimental): A Bruton Tyrosine Kinase Inhibitor
  Interventions: Drug: ibrutinib

INTERVENTIONS:
Drug: ofatumumab — The ofatumumab (IV) dosage and schedule is 12 doses administered over 24 weeks or until disease progression, unacceptable toxicity.
  Week 1: 300 mg initial dose Week 2 through 8: 2,000 mg (once weekly) Week 12, 16, 20 and 24: 2,000 mg (every 4 weeks)
  Arms: Ofatumumab (Arm A)
Drug: ibrutinib — ibrutinib 420 mg (3 x 140-mg capsules) will be administered orally once daily until disease progression or unacceptable toxicity
  Arms: ibrutinib (Arm B)

SUMMARY:
The purpose of the study is to evaluate whether treatment with ibrutinib as a monotherapy results in a clinically significant improvement in progression free survival (PFS) as compared to treatment with ofatumumab in patients with relapsed or refractory Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL)

DETAILED DESCRIPTION:
Study PCYC-1112-CA is a randomized, multicenter, open-label, phase 3 study of the Bruton's Tyrosine Kinase (BTK) inhibitor Ibrutinib (PCI-32765) versus Ofatumumab in patients with Relapsed or Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma.

Patients randomized to the ofatumumab arm may be considered to receive next subsequent therapy with ibrutinib.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of 0-1.
* Diagnosis of CLL or SLL that meets IWCLL 2008 criteria.
* Active disease meeting at least 1 of the IWCLL 2008 criteria for requiring treatment.
* Must have received at least one prior therapy for CLL/SLL.
* Considered not appropriate for treatment or retreatment with purine analog based therapy.
* Measurable nodal disease by CT.
* Patients must be able to receive outpatient treatment and laboratory monitoring at the institution that administers study drug for the entire study.

Exclusion Criteria:

* Known CNS lymphoma or leukemia.
* No documentation of cytogenetic and/or FISH in patient records prior to first dose of study drug.
* Any history of Richter's transformation or prolymphocytic leukemia.
* Uncontrolled Autoimmune Hemolytic Anemia (AIHA) or idiopathic thrombocytopenia purpura (ITP).
* Prior exposure to ofatumumab or to ibrutinib.
* Prior autologous transplant within 6 months prior to first dose of study drug.
* Prior allogeneic stem cell transplant within 6 months or with any evidence of active graft versus host disease or requirement for immunosuppressants within 28 days prior to first dose of study drug.
* History of prior malignancy, with the exception of certain skin cancers and malignancies treated with curative intent and with no evidence of active disease for more than 3 years.
* Serologic status reflecting active hepatitis B or C infection.
* Unable to swallow capsules or disease significantly affecting gastrointestinal function.
* Uncontrolled active systemic fungal, bacterial, viral, or other infection.
* History of stroke or intracranial hemorrhage within 6 months prior to the first dose of study drug.
* Requires anticoagulation with warfarin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2018-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anita Szoke, MD, Study Director — Pharmacyclics LLC.
Locations (76):
- United States (25):
  - Site #408, La Jolla, California
  - Site #377, Los Angeles, California
  - Site #403, Santa Maria, California
  - Site #038, Stanford, California
  - Site #411, Norwalk, Connecticut
  - Site #107, Marietta, Georgia
  - Site # 379, Evansville, Indiana
  - Site # 390, Boston, Massachusetts
  - Site # 391, Boston, Massachusetts
  - Site # 349, Boston, Massachusetts
  - Site # 130, Detroit, Michigan
  - Site # 406, Rochester, Minnesota
  - Site # 059, New Brunswick, New Jersey
  - Site # 350, New Hyde Park, New York
  - Site # 200, New York, New York
  - Site # 127, Rochester, New York
  - Site # 197, Cincinnati, Ohio
  - Site # 217, Columbus, Ohio
  - Site # 402, Philadelphia, Pennsylvania
  - Site # 396, Greenville, South Carolina
  - Site # 410, Nashville, Tennessee
  - Site # 032, Houston, Texas
  - Site # 381, Laredo, Texas
  - Site # 210, Charlottesville, Virginia
  - Site # 404, Seattle, Washington
- Australia (5):
  - Site # 500, St Leonards, New South Wales
  - Site # 503, Brisbane, Queensland
  - Site # 199, East Melbourne, Victoria
  - Site # 501, Fitzroy, Victoria
  - Site # 502, Nedlands, Western Australia
- Austria (6):
  - Site # 509, Graz
  - Site # 508, Linz
  - Site # 504, Salzburg
  - Site # 505, Vienna
  - Site # 506, Wein
  - Site # 507, Wels
- Site # 393, Antwerp, Belgium
- France (9):
  - Site # 519, Argenteuil
  - Site # 511, Bobigny
  - Site # 515, Bordeaux
  - Site # 516, Caen
  - Site # 513, Clermont-Ferrand
  - Site # 510, Marseille
  - Site # 520, Nantes
  - Site # 518, Rennes
  - Site # 517, Vandœuvre-lès-Nancy
- Ireland (3):
  - Site # 570, Dublin
  - Site # 528, Dublin
  - Site # 096, Galway
- Italy (5):
  - Site # 522, Milan
  - Site # 523, Milan
  - Site # 526, Milan
  - Site # 524, Modena
  - Site # 527, Padua
- Poland (2):
  - Site # 529, Gdansk
  - Site # 531, Lodz
- Spain (8):
  - Site # 539, A Coruña
  - Site # 535, Barcelona
  - Site # 534, Barcelona
  - Site # 533, Barcelona
  - Site # 540, Madrid
  - Site # 537, Madrid
  - Site # 536, Madrid
  - Site # 538, Pamplona
- United Kingdom (12):
  - Site # 549, Colchester, Essex
  - Site # 543, Sutton, Surrey
  - Site # 551, Bournemouth
  - Site # 553, Canterbury
  - Site # 546, Cardiff
  - Site # 554, Headington
  - Site # 550, Leeds
  - Site # 552, Liverpool
  - Site # 544, London
  - Site # 548, Nottingham
  - Site # 545, Southampton
  - Site # 541, Withington

REFERENCES:
- [Derived] Abuhelwa AY, Almansour SA, Brown JR, Al-Shamsi HO, Abuhelwa Z, Kharaba Z, Bustanji Y, Semreen MH, Ali S, Alhuraiji A, McKinnon RA, Sorich MJ, Alzoubi KH, Hopkins AM. Statin use and survival in CLL/SLL treated with ibrutinib: pooled analysis of 4 randomized controlled trials. Blood Adv. 2025 Jul 22;9(14):3566-3575. doi: 10.1182/bloodadvances.2024015287. PMID 40266025
- [Derived] Munir T, Brown JR, O'Brien S, Barrientos JC, Barr PM, Reddy NM, Coutre S, Tam CS, Mulligan SP, Jaeger U, Kipps TJ, Moreno C, Montillo M, Burger JA, Byrd JC, Hillmen P, Dai S, Szoke A, Dean JP, Woyach JA. Final analysis from RESONATE: Up to six years of follow-up on ibrutinib in patients with previously treated chronic lymphocytic leukemia or small lymphocytic lymphoma. Am J Hematol. 2019 Dec;94(12):1353-1363. doi: 10.1002/ajh.25638. Epub 2019 Oct 13. PMID 31512258
- [Derived] Coutre SE, Byrd JC, Hillmen P, Barrientos JC, Barr PM, Devereux S, Robak T, Kipps TJ, Schuh A, Moreno C, Furman RR, Burger JA, O'Dwyer M, Ghia P, Valentino R, Chang S, Dean JP, James DF, O'Brien SM. Long-term safety of single-agent ibrutinib in patients with chronic lymphocytic leukemia in 3 pivotal studies. Blood Adv. 2019 Jun 25;3(12):1799-1807. doi: 10.1182/bloodadvances.2018028761. PMID 31196847
- [Derived] Byrd JC, Hillmen P, O'Brien S, Barrientos JC, Reddy NM, Coutre S, Tam CS, Mulligan SP, Jaeger U, Barr PM, Furman RR, Kipps TJ, Thornton P, Moreno C, Montillo M, Pagel JM, Burger JA, Woyach JA, Dai S, Vezan R, James DF, Brown JR. Long-term follow-up of the RESONATE phase 3 trial of ibrutinib vs ofatumumab. Blood. 2019 May 9;133(19):2031-2042. doi: 10.1182/blood-2018-08-870238. Epub 2019 Mar 6. PMID 30842083
- [Derived] O'Brien SM, Jaglowski S, Byrd JC, Bannerji R, Blum KA, Fox CP, Furman RR, Hillmen P, Kipps TJ, Montillo M, Sharman J, Suzuki S, James DF, Chu AD, Coutre SE. Prognostic Factors for Complete Response to Ibrutinib in Patients With Chronic Lymphocytic Leukemia: A Pooled Analysis of 2 Clinical Trials. JAMA Oncol. 2018 May 1;4(5):712-716. doi: 10.1001/jamaoncol.2017.5604. PMID 29470582
- [Derived] Brown JR, Moslehi J, O'Brien S, Ghia P, Hillmen P, Cymbalista F, Shanafelt TD, Fraser G, Rule S, Kipps TJ, Coutre S, Dilhuydy MS, Cramer P, Tedeschi A, Jaeger U, Dreyling M, Byrd JC, Howes A, Todd M, Vermeulen J, James DF, Clow F, Styles L, Valentino R, Wildgust M, Mahler M, Burger JA. Characterization of atrial fibrillation adverse events reported in ibrutinib randomized controlled registration trials. Haematologica. 2017 Oct;102(10):1796-1805. doi: 10.3324/haematol.2017.171041. Epub 2017 Jul 27. PMID 28751558
- [Derived] Barr PM, Brown JR, Hillmen P, O'Brien S, Barrientos JC, Reddy NM, Coutre S, Mulligan SP, Jaeger U, Furman RR, Cymbalista F, Montillo M, Dearden C, Robak T, Moreno C, Pagel JM, Burger JA, Suzuki S, Sukbuntherng J, Cole G, James DF, Byrd JC. Impact of ibrutinib dose adherence on therapeutic efficacy in patients with previously treated CLL/SLL. Blood. 2017 May 11;129(19):2612-2615. doi: 10.1182/blood-2016-12-737346. Epub 2017 Apr 3. PMID 28373262
- [Derived] Maddocks KJ, Ruppert AS, Lozanski G, Heerema NA, Zhao W, Abruzzo L, Lozanski A, Davis M, Gordon A, Smith LL, Mantel R, Jones JA, Flynn JM, Jaglowski SM, Andritsos LA, Awan F, Blum KA, Grever MR, Johnson AJ, Byrd JC, Woyach JA. Etiology of Ibrutinib Therapy Discontinuation and Outcomes in Patients With Chronic Lymphocytic Leukemia. JAMA Oncol. 2015 Apr;1(1):80-7. doi: 10.1001/jamaoncol.2014.218. PMID 26182309
- [Derived] Byrd JC, Brown JR, O'Brien S, Barrientos JC, Kay NE, Reddy NM, Coutre S, Tam CS, Mulligan SP, Jaeger U, Devereux S, Barr PM, Furman RR, Kipps TJ, Cymbalista F, Pocock C, Thornton P, Caligaris-Cappio F, Robak T, Delgado J, Schuster SJ, Montillo M, Schuh A, de Vos S, Gill D, Bloor A, Dearden C, Moreno C, Jones JJ, Chu AD, Fardis M, McGreivy J, Clow F, James DF, Hillmen P; RESONATE Investigators. Ibrutinib versus ofatumumab in previously treated chronic lymphoid leukemia. N Engl J Med. 2014 Jul 17;371(3):213-23. doi: 10.1056/NEJMoa1400376. Epub 2014 May 31. PMID 24881631

RESULTS

PARTICIPANT FLOW:
Groups:
- Ofatumumab (Arm A): An anti-CD20 monoclonal antibody
  ofatumumab: The ofatumumab (IV) dosage and schedule is 12 doses administered over 24 weeks or until disease progression, unacceptable toxicity.
  Week 1: 300 mg initial dose Week 2 through 8: 2,000 mg (once weekly) Week 12, 16, 20 and 24: 2,000 mg (every 4 weeks)
Period: Overall Study
Arm/Group | Ofatumumab (Arm A) | Ibrutinib (Arm B)
Started | 196 | 195
Completed | 196 | 195
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ofatumumab (Arm A) | Ibrutinib (Arm B) | Total
Number analyzed (Participants) | 196 | 195 | 391
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 77 | 152
  >=65 years | 121 | 118 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (8.88) | 66.1 (10.15) | 66.5 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 66 | 125
  Male | 137 | 129 | 266

OUTCOME MEASURES:

1. Primary Outcome: PFS (Progression Free Survival) by Independent Review Committee (IRC), Limited to the Time of Primary Analysis 06 November 2013
Description: The primary objective of this study was to evaluate the efficacy of ibrutinib compared to ofatumumab based on independent review committee (IRC) assessment of progression-free survival (PFS) according to 2008 IWCLL guidelines.
Time Frame: Analysis was conducted after observing approximately 117 PFS events, which occurred about 18 months after the first subject was enrolled.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ofatumumab (Arm A) | Ibrutinib (Arm B)
Number analyzed (Participants) | 196 | 195
months | 8.1 [7.2 to 8.3] | NA [NA to NA] — IBR: Median PFS was not reached so 95% CI for median PFS is not applicable.
Statistical Analysis 1: Comparison: Ofatumumab (Arm A); Test type: Superiority; p < 0.0001, Log Rank

2. Secondary Outcome: Overall Response Rate (ORR) by Independent Review Committee (IRC)
Description: Overall Response Rate per the IWCLL 2008 criteria as assessed by IRC, limited to the time of primary analysis 06 November 2013
Time Frame: About 18 months after the first subject was enrolled
Measure: Number; unit: percentage of participants
Arm/Group | Ofatumumab (Arm A) | Ibrutinib (Arm B)
Number analyzed (Participants) | 196 | 195
percentage of participants | 4.1 | 42.6
Statistical Analysis 1: Comparison: Ofatumumab (Arm A); Test type: Superiority; p < .0001, Fisher Exact

3. Secondary Outcome: OS (Overall Survival)
Description: OS analysis was conducted at the time of study closure, with no adjustment for crossover from the ofatumumab arm to the ibrutinib arm
Time Frame: OS analysis was conducted at the time of study closure, including up to 6 years of study follow-up
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ofatumumab (Arm A) | Ibrutinib (Arm B)
Number analyzed (Participants) | 196 | 195
months | 65.1 [50.6 to NA] — OFA: Upper limit of 95% CI for median OS is not estimable due to sparse events in the data / insufficient number of participants with events. | 67.7 [61.0 to NA] — IBR: Upper limit of 95% CI for median OS is not estimable due to sparse events in the data / insufficient number of participants with events.
Statistical Analysis 1: Comparison: Ofatumumab (Arm A); Test type: Superiority or Other; p = 0.1653, Log Rank

4. Secondary Outcome: Rate of Sustained Hemoglobin and Platelet Improvement
Description: Proportion of subjects with hemoglobin (HgB) increase >=20 g/L and platelet (PLT) increase >=50% over baseline continuously for >=56 days without blood transfusions or growth factors.
Time Frame: From study initiation to study closure, including up to 6 years of study follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Ofatumumab (Arm A) | Ibrutinib (Arm B)
Number analyzed (Participants) | 196 | 195
percentage of participants
  Hgb Improvement in patient with baseline anemia | 32.6 | 69.7
  Platelet improvement in baseline thrombocytopenia | 9.4 | 78.4

5. Other Pre Specified Outcome: Progression Free Survival (PFS) by Investigator With up to 6 Years of Study Follow-up
Description: Long-Term Progression Free Survival as assessed by the investigator with up to 6 years of study follow-up
Time Frame: From study initiation to study closure, including up to 6 years of study follow-up
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ofatumumab (Arm A) | Ibrutinib (Arm B)
Number analyzed (Participants) | 196 | 195
months | 8.1 [7.79 to 8.25] | 44.1 [38.47 to 56.18]

6. Other Pre Specified Outcome: Overall Response Rate (ORR) by Investigator
Description: Overall response per the IWCLL 2008 criteria as assessed by Investigator with up to 6 years of study follow-up
Time Frame: From study initiation to study closure, including up to 6 years of study follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Ofatumumab (Arm A) | Ibrutinib (Arm B)
Number analyzed (Participants) | 196 | 195
percentage of participants | 22.4 | 87.7

ADVERSE EVENTS:
Time Frame: From first dose of study drug to within 30 days of last dose.
Description: 196 subjects were randomized to the Ofa arm with 191 received drug thus 5 patients were not included in the number of participants at risk.
Arm/Group | Ofatumumab (Arm A) | Ibrutinib (Arm B)
All-Cause Mortality (participants affected / at risk) | 16/191 | 24/195
Serious Adverse Events (participants affected / at risk) | 59/191 | 141/195
Other Adverse Events (participants affected / at risk) | 185/191 | 194/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab (Arm A) (N=191) | Ibrutinib (Arm B) (N=195)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 | 7
Anaemia (Blood and lymphatic system disorders) | 4 | 5
Neutropenia (Blood and lymphatic system disorders) | 2 | 4
Spontaneous Haematoma (Blood and lymphatic system disorders) | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Autoimmune Haemolytic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Haemolytic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Methaemoglobinaemia (Blood and lymphatic system disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 11
Cardiac Failure Congestive (Cardiac disorders) | 0 | 3
Atrioventricular Block (Cardiac disorders) | 0 | 2
Cardiac Failure (Cardiac disorders) | 1 | 2
Myocardial infarction (Cardiac disorders) | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina Pectoris (Cardiac disorders) | 0 | 1
Aortic Valve Disease (Cardiac disorders) | 0 | 1
Atrial Tachycardia (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 1
Myocardial Ischaemia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pericardial Effusion (Cardiac disorders) | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 1 | 1
Sinus Tachycardia (Cardiac disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Vitreous Haemorrhage (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 6
Vomiting (Gastrointestinal disorders) | 0 | 5
Abdominal Pain (Gastrointestinal disorders) | 1 | 4
Nausea (Gastrointestinal disorders) | 0 | 3
Umbilical Hernia (Gastrointestinal disorders) | 0 | 2
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1
Anorectal Discomfort (Gastrointestinal disorders) | 0 | 1
Duodenal Perforation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Mucous stools (Gastrointestinal disorders) | 0 | 1
Oesophageal Obstruction (Gastrointestinal disorders) | 0 | 1
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Poor Dental Condition (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Malabsorption (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 4 | 15
Non-Cardiac Chest Pain (General disorders) | 0 | 3
Malaise (General disorders) | 0 | 2
Sudden Death (General disorders) | 0 | 2
Asthenia (General disorders) | 0 | 1
Catheter Site Pain (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Cyst (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
General Physical Health Deterioration (General disorders) | 0 | 1
Influenza Like Illness (General disorders) | 0 | 1
Injection Site Extravasation (General disorders) | 0 | 1
Effusion (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1
Anaphylactic Shock (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 12 | 42
Urinary Tract Infection (Infections and infestations) | 0 | 9
Cellulitis (Infections and infestations) | 1 | 8
Sepsis (Infections and infestations) | 2 | 8
Lung Infection (Infections and infestations) | 0 | 7
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 4
Lower Respiratory Tract Infection (Infections and infestations) | 2 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 4
Infection (Infections and infestations) | 1 | 3
Aspergillus Infection (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 2 | 2
Bronchopulmonary Aspergillosis (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 2
Gastroenteritis Viral (Infections and infestations) | 0 | 2
Herpes Zoster (Infections and infestations) | 1 | 2
Influenza (Infections and infestations) | 2 | 2
Neutropenic Sepsis (Infections and infestations) | 2 | 2
Pneumocystis Jirovecii Ppneumonia (Infections and infestations) | 1 | 2
Pneumonia Pseudomonal (Infections and infestations) | 1 | 2
Pneumonia Staphylococcal (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 0 | 2
Urosepsis (Infections and infestations) | 0 | 2
Bacteraemia (Infections and infestations) | 2 | 1
Bacterial Infection (Infections and infestations) | 0 | 1
Bacteroides Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis Bacterial (Infections and infestations) | 0 | 1
Campylobacter Gastroenteritis (Infections and infestations) | 0 | 1
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1
Clostridium Difficile Infection (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 0 | 1
Enterococcal Iinfection (Infections and infestations) | 0 | 1
Enterococcal Sepsis (Infections and infestations) | 0 | 1
Enterocolitis Infectious (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 1
Gastrointestinal Infection (Infections and infestations) | 0 | 1
H1N1 Influenza (Infections and infestations) | 0 | 1
Haemophilus Bacteraemia (Infections and infestations) | 0 | 1
Haemophilus Infection (Infections and infestations) | 0 | 1
Haemophilus Sepsis (Infections and infestations) | 0 | 1
Herpes Virus Infection (Infections and infestations) | 0 | 1
Impetigo (Infections and infestations) | 0 | 1
Infective Exacerbation of Bronchiectasis (Infections and infestations) | 0 | 1
Intervertebral Discitis (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection Bacterial (Infections and infestations) | 0 | 1
Lymph Gland Infection (Infections and infestations) | 0 | 1
Meningitis Pneumococcal (Infections and infestations) | 0 | 1
Mycobacterium Avium Complex Infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Otitis Externa (Infections and infestations) | 0 | 1
Otitis Media (Infections and infestations) | 0 | 1
Parainfluenzae Virus Infection (Infections and infestations) | 0 | 1
Pneumococcal Sepsis (Infections and infestations) | 0 | 1
Pneumocystis Jirovecii Infection (Infections and infestations) | 0 | 1
Pneumonia Bacterial (Infections and infestations) | 1 | 1
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 1
Pseudomonal Sepsis (Infections and infestations) | 0 | 1
Pseudomonas Infection (Infections and infestations) | 2 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 2 | 1
Rhinovirus Infection (Infections and infestations) | 0 | 1
Septic Shock (Infections and infestations) | 1 | 1
Staphylococcal Sepsis (Infections and infestations) | 0 | 1
Staphylococcal Skin Infection (Infections and infestations) | 0 | 1
Tonsillitis Fungal (Infections and infestations) | 0 | 1
Tooth Infection (Infections and infestations) | 0 | 1
Urethritis (Infections and infestations) | 0 | 1
Urinary Tract Infection Pseudomonal (Infections and infestations) | 0 | 1
Viral Pharyngitis (Infections and infestations) | 0 | 1
Abscess Limb (Infections and infestations) | 1 | 0
Anal Infection (Infections and infestations) | 1 | 0
Breast Cellulitis (Infections and infestations) | 1 | 0
Febrile Infection (Infections and infestations) | 1 | 0
Herpes Simplex (Infections and infestations) | 1 | 0
Infectious Pleural Effusion (Infections and infestations) | 1 | 0
Lung Infection Pseudomonal (Infections and infestations) | 1 | 0
Nocardiosis (Infections and infestations) | 1 | 0
Ophthalmic Herpes Zoster (Infections and infestations) | 1 | 0
Pneumonia Mycoplasmal (Infections and infestations) | 1 | 0
Sepsis Syndrome (Infections and infestations) | 1 | 0
Stenotrophomonas Infection (Infections and infestations) | 2 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 6
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 4
Fall (Injury, poisoning and procedural complications) | 0 | 2
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 2
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 1
Brain Contusion (Injury, poisoning and procedural complications) | 0 | 1
Burns Third Degree (Injury, poisoning and procedural complications) | 0 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Multiple Fractures (Injury, poisoning and procedural complications) | 1 | 1
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 1
Subarachnoid Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Subarachnoid Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 1
Traumatic Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 2 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 0
Immunoglobulins Decreased (Investigations) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 1
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Richter's Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bone Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Desmoid Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Histiocytic Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraductal Papillary Mucinous Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous Cell Carcinoma of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour Flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Seizure (Nervous system disorders) | 0 | 3
Cerebrovascular Accident (Nervous system disorders) | 0 | 2
Transient Ischaemic Attack (Nervous system disorders) | 0 | 2
Cerebral Haemorrhage (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Mental Status Changes (Psychiatric disorders) | 0 | 3
Depression (Psychiatric disorders) | 0 | 1
Hallucination, Visual (Psychiatric disorders) | 0 | 1
Mania (Psychiatric disorders) | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 0
Major Depression (Psychiatric disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 2 | 4
Haematuria (Renal and urinary disorders) | 0 | 2
Urinary Retention (Renal and urinary disorders) | 0 | 2
Calculus Bladder (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 1 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Pyoderma Gangrenosum (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Aneurysm (Vascular disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab (Arm A) (N=191) | Ibrutinib (Arm B) (N=195)
Anaemia (Blood and lymphatic system disorders) | 32 | 62
Neutropenia (Blood and lymphatic system disorders) | 25 | 60
Increased Tendency to Bruise (Blood and lymphatic system disorders) | 4 | 45
Thrombocytopenia (Blood and lymphatic system disorders) | 22 | 45
Lymphocytosis (Blood and lymphatic system disorders) | 5 | 10
Atrial Fibrillation (Cardiac disorders) | 0 | 19
Dry Eye (Eye disorders) | 10 | 33
Vision Blurred (Eye disorders) | 6 | 30
Lacrimation Increased (Eye disorders) | 5 | 27
Cataract (Eye disorders) | 2 | 26
Visual Acuity Reduced (Eye disorders) | 1 | 19
Eye Irritation (Eye disorders) | 3 | 17
Eye Pain (Eye disorders) | 5 | 15
Photophobia (Eye disorders) | 4 | 14
Vitreous Floaters (Eye disorders) | 3 | 14
Diarrhoea (Gastrointestinal disorders) | 33 | 120
Nausea (Gastrointestinal disorders) | 38 | 69
Constipation (Gastrointestinal disorders) | 19 | 45
Vomiting (Gastrointestinal disorders) | 11 | 39
Abdominal Pain (Gastrointestinal disorders) | 19 | 30
Stomatitis (Gastrointestinal disorders) | 5 | 30
Dyspepsia (Gastrointestinal disorders) | 6 | 22
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3 | 21
Dry Mouth (Gastrointestinal disorders) | 1 | 19
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 16
Flatulence (Gastrointestinal disorders) | 2 | 10
Haemorrhoids (Gastrointestinal disorders) | 3 | 10
Fatigue (General disorders) | 57 | 82
Pyrexia (General disorders) | 27 | 66
Oedema Peripheral (General disorders) | 16 | 46
Asthenia (General disorders) | 8 | 22
Chills (General disorders) | 6 | 16
Influenza Like Illness (General disorders) | 5 | 16
Malaise (General disorders) | 1 | 10
Upper Respiratory Tract Infection (Infections and infestations) | 17 | 77
Sinusitis (Infections and infestations) | 12 | 50
Urinary Tract Infection (Infections and infestations) | 10 | 46
Bronchitis (Infections and infestations) | 2 | 28
Nasopharyngitis (Infections and infestations) | 7 | 22
Conjunctivitis (Infections and infestations) | 2 | 21
Pneumonia (Infections and infestations) | 3 | 21
Cellulitis (Infections and infestations) | 3 | 15
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 15
Herpes Zoster (Infections and infestations) | 3 | 14
Ear Infection (Infections and infestations) | 2 | 13
Folliculitis (Infections and infestations) | 0 | 10
Contusion (Injury, poisoning and procedural complications) | 6 | 38
Fall (Injury, poisoning and procedural complications) | 1 | 18
Traumatic Haematoma (Injury, poisoning and procedural complications) | 0 | 12
Infusion Related Reaction (Injury, poisoning and procedural complications) | 64 | 0
Weight Decreased (Investigations) | 11 | 25
Blood Creatinine Increased (Investigations) | 0 | 12
Platelet Count Decreased (Investigations) | 0 | 11
Weight Increased (Investigations) | 0 | 11
Decreased Appetite (Metabolism and nutrition disorders) | 16 | 32
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 22
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 22
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 16
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 53
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 16 | 46
Back Pain (Musculoskeletal and connective tissue disorders) | 14 | 39
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 9 | 29
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 24
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 9 | 20
Bone Pain (Musculoskeletal and connective tissue disorders) | 3 | 10
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3 | 10
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 10
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 18
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 13
Headache (Nervous system disorders) | 12 | 41
Dizziness (Nervous system disorders) | 10 | 33
Peripheral Sensory Neuropathy (Nervous system disorders) | 26 | 22
Paraesthesia (Nervous system disorders) | 10 | 14
Anxiety (Psychiatric disorders) | 9 | 18
Depression (Psychiatric disorders) | 3 | 17
Insomnia (Psychiatric disorders) | 16 | 17
Confusional State (Psychiatric disorders) | 4 | 11
Pollakiuria (Renal and urinary disorders) | 3 | 19
Dysuria (Renal and urinary disorders) | 1 | 12
Haematuria (Renal and urinary disorders) | 2 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 43 | 78
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 33
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 32
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 30
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 19
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 17
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 14
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 14
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 10
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 28
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 7 | 26
Night Sweats (Skin and subcutaneous tissue disorders) | 23 | 24
Skin Lesion (Skin and subcutaneous tissue disorders) | 5 | 24
Rash Erythematous (Skin and subcutaneous tissue disorders) | 9 | 20
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 19
Rash (Skin and subcutaneous tissue disorders) | 7 | 19
Dry Skin (Skin and subcutaneous tissue disorders) | 3 | 18
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 5 | 16
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 12
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 12
Blood Blister (Skin and subcutaneous tissue disorders) | 1 | 10
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 10
Hypertension (Vascular disorders) | 4 | 40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-09-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT01578707/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT01578707/SAP_001.pdf